CLINICAL TRIAL: NCT05690334
Title: Up-and-Down Determination of Different Crystalloid Coload Volumes on the 90% Effective Dose of Prophylactic Norepinephrine Infusions for Preventing Postspinal Anesthesia Hypotension During Cesarean Section
Brief Title: Different Crystalloid Coload Volumes on the 90% ED of Norepinephrine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Yi Chen-2023-2
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Adverse Effect
Keywords: Norepinephrine; Postspinal anesthesia hypotension; Coload; Cesarean section
MeSH Terms: interventions — Crystalloid Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Experimental): No fluid coload was given. An initial infusion dose of prophylactic norepinephrine simultaneous with spinal anesthesia
  Interventions: Drug: Crystalloid - 0 ml/kg
- Crystalloid - 5 ml/kg (Experimental): 5 ml/kg crystalloid coload combined with an initial infusion dose of prophylactic norepinephrine simultaneous with spinal anesthesia.
  Interventions: Drug: Crystalloid - 5 ml/kg
- Crystalloid - 10 ml/kg (Experimental): 10 ml/kg crystalloid coload combined with an initial infusion dose of prophylactic norepinephrine simultaneous with spinal anesthesia.
  Interventions: Drug: Crystalloid - 10 ml/kg

INTERVENTIONS:
Drug: Crystalloid - 0 ml/kg — No fluid coload was given. An initial infusion dose of prophylactic norepinephrine (0.025 ug/kg/min) simultaneous with spinal anesthesia. The dose administered to subsequent patients varied by increments or decrements of 0.005 ug/kg/min of prophylactic norepinephrine according to the responses of previous patients according to the up-down sequential allocation.
  Other Names: Crystalloid
  Arms: Control group
Drug: Crystalloid - 5 ml/kg — 5 ml/kg crystalloid coload combined with an initial infusion dose of prophylactic norepinephrine (0.025 ug/kg/min) simultaneous with spinal anesthesia. The dose administered to subsequent patients varied by increments or decrements of 0.005 ug/kg/min of prophylactic norepinephrine according to the responses of previous patients according to the up-down sequential allocation.
  Other Names: Crystalloid
  Arms: Crystalloid - 5 ml/kg
Drug: Crystalloid - 10 ml/kg — 10 ml/kg crystalloid coload combined with an initial infusion dose of prophylactic norepinephrine (0.025 ug/kg/min) simultaneous with spinal anesthesia. The dose administered to subsequent patients varied by increments or decrements of 0.005 ug/kg/min of prophylactic norepinephrine according to the responses of previous patients according to the up-down sequential allocation.
  Other Names: Crystalloid
  Arms: Crystalloid - 10 ml/kg

SUMMARY:
The purpose of this study is to investigate the effect of different crystalloid coload volumes on the 90% effective dose of prophylactic norepinephrine infusions for preventing postspinal anesthesia hypotension during cesarean section.

DETAILED DESCRIPTION:
Post-spinal anesthesia hypotension is a frequent complication during spinal anesthesia for cesarean section. The incidence of post-spinal anesthesia hypotension is as high as 62.1-89.7% if prophylactic measures are not taken. Coload has been highly demonstrated for prevention and/or treatment of post-spinal anesthesia hypotension. In addition, there's some evidence that prophylactic infusion of norepinephrine could effectively reduce the incidence of post-spinal anesthesia hypotension in parturients undergoing cesarean section. The purpose of this study is to investigate the effect of different crystalloid coload volumes on the 90% effective dose of norepinephrine infusion prophylaxis for hypotension during spinal anesthesia for cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years
* Primipara or multipara
* Singleton pregnancy ≥37 weeks
* American Society of Anesthesiologists physical status classification I to II
* Scheduled for cesarean section under spinal anesthesia

Exclusion Criteria:

* Body height < 150 cm
* Body weight > 100 kg or body mass index (BMI) ≥ 40 kg/m2
* Eclampsia or chronic hypertension or baseline blood pressure ≥180 mmHg
* Hemoglobin < 7g/dl
* Fetal distress, or known fetal developmental anomaly

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
ED50 and ED90 | 1-15 minutes after spinal anesthesia
  The dose of prophylactic norepinephrine that would be effective in preventing postspinal anesthesia hypotension in 50% (effective dose, ED 50) and 90% (ED90) of patients

SECONDARY OUTCOMES:
The incidence of post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 80% of the baseline
The incidence of severe post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 60% of the baseline
The incidence of bradycardia | 1-15 minutes after spinal anesthesia
  Heart rate < 60 beats/min
The incidence of nausea and vomiting | 1-15 minutes after spinal anesthesia
  Presence of nausea and vomiting in patients after spinal anesthesia
The incidence of hypertension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) >120% of the baseline
pH | Immediately after delivery
  From umbilical arterial blood gases
Partial pressure of oxygen (PO2) | Immediately after delivery
  From umbilical arterial blood gases
Base excess (BE) | Immediately after delivery
  From umbilical arterial blood gases
APGAR score | 1 minute after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration
APGAR score | 5 minute after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration

CONTACTS AND LOCATIONS:
Overall Officials: Yi Chen, M.D., Study Chair — General Hospital of Ningxia Medical University; Xiangsheng Xiong, M.D., Study Chair — The Fifth People's Hospital of Huaian
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China